CLINICAL TRIAL: NCT02650258
Title: Cadence and Intensity Across the Adult Lifespan
Acronym: CADENCE-Adults
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Sponsor
Other Study IDs: 1R01AG049024 (NIH)
Record Dates: First submitted 2015-12-24; First posted 2016-01-08 (Estimated); Last update posted 2022-12-06 (Actual); Status verified 2020-10

CONDITIONS: Aging; Walking; Motor Activity; Activities of Daily Living
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Young Adult: 80 Adults 21-40 years of age: 10 Male and 10 Female in each 5 year increment (21-25, 26-30, 31-35, 36-40).
  Interventions: Behavioral: treadmill walking
- Middle Aged Adults: 80 Adults 41-60 years of age: 10 Male and 10 Female in each 5 year increment (41-45, 46-50, 51-55, 56-60).
  Interventions: Behavioral: treadmill walking
- Older Adults: 100 Adults 61-85 years of age: 10 Male and 10 Female in each 5 year increment (61-65, 66-69, 70-75, 76-80, 81-85).
  Interventions: Behavioral: treadmill walking

INTERVENTIONS:
Behavioral: treadmill walking — all participants walking at increasing speeds on a treadmill

SUMMARY:
The purpose of this study is to determine and link cadence (the number of steps taken in a minute) to the intensity of physical activity (e.g. low-, moderate- and vigorous-intensity) in adults (21-85 years old). The investigators anticipate that cadence will be a good indicator of exercise intensity. Identifying how cadence relates to activity intensity will allow for physical activity guidelines to be communicated to the public in a manner that is more accessible to the lay person.

DETAILED DESCRIPTION:
There will be up to two lab visits for CADENCE-ADULTS participants, all of which will be completed in the Physical Activity and Health Lab at University of Massachusetts Amherst. Participation will include: orientation to the experiment, consent, physical examination and testing. The entire research protocol will last between 3.5-4.5 hrs.

For all participants the first visit will consist of an orientation to the project, screening, informed consent, physical exam and ECG (if necessary, see below), as well as the graded treadmill walking protocol.

Pre-visit:

Prior to coming to the laboratory participants will undergo a phone screening in order to identify interest, outline basic inclusion/exclusion criteria and give a brief description of the study protocol. If interested participants will be scheduled for their first visit and be given the instruction to arrive at the laboratory having observed at least a 4-hour fast.

The reason for required fast is that metabolic responses to exercise are affected by food intake. By fasting for 4 hrs prior to the exercise testing window the investigators insure standardization of metabolic responses to exercise.

Orientation:

Participants will be taken through a slide orientation session where all aspects of the study will be covered. This slide set has both written and pictorial descriptions of the different phases of the experiment, eligibility criteria, participant rights, compensation and confidentially. At this time participants have the opportunity to ask any questions of the experimenters that they would like.

Consent:

If after being presented with the orientation information a person would like to enroll in the study they will be given the informed consent document. They will be given ample opportunity to read through the document and decide if they would like to sign the paper and enroll in the study.

Pre-testing screening:

Once the consent paperwork is signed participants will have their height, seating height, body weight, body fat percentage, BMI, and waist circumference taken. Questions will also be asked to ascertain date of birth, gender and race/ethnicity. Participants will then be taken through a series of screening questionnaires to assess cardio-metabolic risk via the the most recent edition of the American College of Sports Medicine (ACSM) Resource for The Health Fitness Specialist and also the American heart Association's (AHA) risk stratification recommendations presented in the same ACSM resource. Risk will be assessed in the following ways:

For participants considered low risk (men 21-44 years of age and women 21-54 years of age, asymptomatic and with ≤ 1 risk factors) no physical examination and resting ECG is necessary prior to enrolling in the study. Those considered at moderate risk (men 45-69 and women 55-69 years of age, asymptomatic with ≥ 2 risk factors) will require the physical examination and resting ECG prior to enrolling in the study. Those considered to be high risk (symptomatic, or with known cardiac, pulmonary or metabolic disease), or found to be at high risk following risk stratification, will require medical supervision during the submaximal treadmill exercise protocol.

All participants who are 61-85 years of age will require a physical examination and resting ECG prior to enrolling.

Physical Exam and ECG:

A physical exam will be conducted by our study staff under the guidance of our medical examiner (Dr. Chipkin) to assess for medical conditions that may interfere with exercise protocol. In addition, this is being performed to ensure participant safety during exercise protocol .

Electrocardiogram (ECG). A 12-lead electrocardiogram will be performed by study staff and reviewed by a clinical exercise specialist (e.g., clinical exercise physiologist) or MD prior to exercise protocol.

All testing will be overseen by trained study staff with an MS or PhD in Exercise Science/Physiology or BS in Kinesiology. These accommodations meet the latest ACSM (10 Edition, Guidelines for Exercise Testing and Prescription) and AHA criteria for exercise protocols.

Experimental Testing:

Immediately prior to exercise testing participants will be outfitted with a number of non-invasive devices to measure/monitor physical activity. Additionally they will be outfitted with a wireless metabolic mask to measure gas exchange for a criterion measure of energy expenditure.

Participants will complete both the treadmill testing and mock free-living activities while physical activity and oxygen uptake are continually and concurrently measured.

Each speed on the treadmill and each free-living activity will be performed for 5 minutes with a 2 minute rest between each activity. Participants will complete each activity at their preferred level of effort.

Treadmill walking:

Participants will then complete a series of walking bouts on a treadmill while their physical activity and oxygen uptake are concurrently assessed. The walking bouts start at 0.5 miles per hour and end at 6 miles per hour (0.5 miles per hour increments). Treadmill testing will be terminated when any of the following criteria are attained: upon any natural tendency to reach out to use the hand rails to steady and/or support themselves, following completion of the fist bout when their heart rate attains 75% of age-predicted maximum heart rate(indicative of having achieved vigorous intensity), participants identify as having a 14/20 or greater level of exertion on a Borg Rate of Perceived Exertion Scale, following completion of first bout when the participant naturally selects to run instead of walk, following completion of a bout at 6.0 mph, or before any of the above criteria, as the participant prefers, reflecting their personal tolerance.

Free-Living Activities:

Participants will rest in chair, watch a portion of a movie while seated in a chair, complete seated computer work, walk up and down a set of stairs, fold laundry while standing, and vacuum the floor. Participant will then complete a continuous walk for 5 minutes at their desired pace. This walk will be completed in a corridor with an electronic gait mat (GaitRite, Inc., USA) covering a portion of the walking course.

Following completion of the testing, participants will be given a small snack and drink and will be monitored to ensure it is safe for them to return to their day.

NIH NIA supplement award R01AG049024-05S1, start date May 2018 -

In addition to the above procedures related to the CADENCE-Adults parent award, participants aged 61-85 may also participate in an optional component of the study related to the supplement award. This will include:

1 week of physical activity monitoring: An additional 7 consecutive days of physical activity monitoring (ActiGraph GT9X and New Lifestyle DigiWalker SW-200). Participants will wear the devices on their waist for 24 hours a day and maintain their usual physical activity levels. They will also be asked to complete a daily physical activity log. Participants will be to complete this within twelve weeks of their final visit to the physical activity and health lab. In addition, they will also be asked a series questions regarding their physical activity history over the past month (CHAMPS questionnaire).

AND Peak aerobic fitness treadmill protocol (modified Balke protocol). Participants will will first walk for a warm-up period of 6 - 10 minutes at a comfortable walking speed. Treadmill speed will then be set to elicit 70-80% of their age-predicted max heart-rate (HRmax), and remain constant for the entirety of the protocol. This speed will be determined based on the speed and heart rate relationship observed during the previous treadmill test (sub-maximal treadmill protocol). Specifically, if 70% of HRmax was reached during the previous test, the peak aerobic fitness test will start at the first speed at which this heart rate threshold was first observed. If the previous test was terminated before 70% of HRmax (e.g., the participant naturally chose to run or achieved a rating perceived exertion consistent with a vigorous intensity), the speed for the peak protocol will be set at 0.5 mph faster than the previous test's termination speed. If the previous test was terminated before 70% of HRmax was reached because the participant: indicated they wished to stop the test, the researchers stopped the test due to safety concerns, they reached for the handrail or became unsteady, or they achieved a systolic blood pressure >200 mmHg or diastolic blood pressure >110 mmHg; then the speed for the peak protocol will be set 0.5 mph slower than the previous termination speed.

Participant will first walk at the pre-determined testing speed for 2 minutes at a grade (incline) of 0%. The grade will then be increased from 0% to 4% after 2-minutes, then to 6% after 4 minutes, and then by 2% every minute thereafter until they indicate that they want to stop (voluntary exhaustion), or earlier for any safety-related reasons. During this testing, the participant will be outfitted with the Oxycon Mobile to assess peak aerobic fitness.

For safety reasons, participants will be required to wear the ECG and BP equipment to monitor their cardiovascular responses during this test. A trained staff member will be on hand to operate this equipment, monitor responses and ensure safety procedures are followed. Our medical investigator, Dr Stuart Chipkin will be on hand to supervise all peak treadmill protocols.

Participants will be required to complete this a minimum of 7 days, and maximum of 12 weeks from the the submaximal treadmil protocol in the parent award.

ELIGIBILITY:
Inclusion Criteria:

* Adults between ages 21-85 years, able to ambulate on a treadmill (self-report)

Exclusion Criteria:

* BMI less than 18.5 or more than 40kg/m^2
* Having smoked tobacco within the past 6 months
* wheelchair bound, or conditions that prevent normal ambulation
* Resting systolic blood pressure > 159 mm HG, or diastolic blood pressure > 99 mm HG
* Hospitalization for mental illness within the past 5 years (for the 41-60 and 61-85 year old cohorts this was change to "within the past 1 year").
* Any condition/medication that may affect heart rate response to exercise testing.
* Previous history of, or clinical symptoms or signs of, cardiovascular disease, stroke or transient ischemic attacks, chest pain, unusual dyspnea during physical activity/exercise, severe ankle swelling, or leg pain while walking.
* Any significant medical condition that may interfere with the study.
* Previous history of musculoskeletal injuries or problems causing severe pain during physical activity or exercise which interferes with daily activities.
* Participant has a pacemaker or other implanted medical device (including metal joint replacements).
* Participant is pregnant.
* Participant is unable to complete all testing (1 or two sessions, based on risk factors) within a maximal two week period.
* Individuals wearing a full beard may need to be excluded from the study, as large amounts of facial hair around the mouth and nose interfere with the seal of the device that measures the air you breath. Because of this we are seeking participants that are clean-shaven or with a beard where areas around the nose and mouth are clean-shaven (e.g. goatee).

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A convenience sample from the surrounding community of male and females 21-85 years will be recruited as participants. Specifically, 10 men and 10 women for each 5-year age-group category (21-25, 26-30, 31-35, etc.) will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2015-12; Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Cadence (steps/min) as assessed by observation (hand tallied counts) of cadence | Cross-sectional data; single time point, throughout study, up to 5 years
  The identification of cadence value cut-points associated with low, moderate and vigorous activity.
Monitor validation (difference in steps/min compared to observation/hand tallied counts) | Cross-sectional data; single time point, throughout study, up to 5 years
  Compare the ability of different activity monitors to accurately measure cadence

CONTACTS AND LOCATIONS:
Overall Officials: Catrine Tudor-Locke, PhD, Principal Investigator — University of North Carolina at Charlotte
Locations (1):
- Walking Research Laboratory, University of North Carolina at Charlotte, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Requests for de-identified individual-level data (including descriptors) collected in CADENCE-Adults and used in publications will be considered and made available to qualified researchers within 2 years of publication of the associated paper. Data sharing agreements will be necessary for access.The CADENCE-Adults data base will be maintained and access ensured by the Physical Activity and Health Laboratory in the Department of Kinesiology at University of Massachusetts Amherst.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Researchers can request supporting information for two years post-publication
Access Criteria: Contact PI

REFERENCES:
- [Background] Tudor-Locke C, Rowe DA. Using cadence to study free-living ambulatory behaviour. Sports Med. 2012 May 1;42(5):381-98. doi: 10.2165/11599170-000000000-00000. PMID 22462794
- [Background] Tudor-Locke C, Sisson SB, Collova T, Lee SM, Swan PD. Pedometer-determined step count guidelines for classifying walking intensity in a young ostensibly healthy population. Can J Appl Physiol. 2005 Dec;30(6):666-76. doi: 10.1139/h05-147. PMID 16485518
- [Background] Tudor-Locke C, Camhi SM, Leonardi C, Johnson WD, Katzmarzyk PT, Earnest CP, Church TS. Patterns of adult stepping cadence in the 2005-2006 NHANES. Prev Med. 2011 Sep;53(3):178-81. doi: 10.1016/j.ypmed.2011.06.004. Epub 2011 Jun 25. PMID 21708187
- [Background] Tudor-Locke C, Han H, Aguiar EJ, Barreira TV, Schuna JM Jr, Kang M, Rowe DA. How fast is fast enough? Walking cadence (steps/min) as a practical estimate of intensity in adults: a narrative review. Br J Sports Med. 2018 Jun;52(12):776-788. doi: 10.1136/bjsports-2017-097628. PMID 29858465
- [Background] Moore CC, McCullough AK, Aguiar EJ, Ducharme SW, Tudor-Locke C. Toward Harmonized Treadmill-Based Validation of Step-Counting Wearable Technologies: A Scoping Review. J Phys Act Health. 2020 Jul 11;17(8):840-852. doi: 10.1123/jpah.2019-0205. Print 2020 Aug 1. PMID 32652514
- [Result] Tudor-Locke C, Aguiar EJ, Han H, Ducharme SW, Schuna JM Jr, Barreira TV, Moore CC, Busa MA, Lim J, Sirard JR, Chipkin SR, Staudenmayer J. Walking cadence (steps/min) and intensity in 21-40 year olds: CADENCE-adults. Int J Behav Nutr Phys Act. 2019 Jan 17;16(1):8. doi: 10.1186/s12966-019-0769-6. PMID 30654810
- [Result] Tudor-Locke C, Ducharme SW, Aguiar EJ, Schuna JM Jr, Barreira TV, Moore CC, Chase CJ, Gould ZR, Amalbert-Birriel MA, Mora-Gonzalez J, Chipkin SR, Staudenmayer J. Walking cadence (steps/min) and intensity in 41 to 60-year-old adults: the CADENCE-adults study. Int J Behav Nutr Phys Act. 2020 Nov 10;17(1):137. doi: 10.1186/s12966-020-01045-z. PMID 33168018
- [Result] Tudor-Locke C, Mora-Gonzalez J, Ducharme SW, Aguiar EJ, Schuna JM Jr, Barreira TV, Moore CC, Chase CJ, Gould ZR, Amalbert-Birriel MA, Chipkin SR, Staudenmayer J. Walking cadence (steps/min) and intensity in 61-85-year-old adults: the CADENCE-Adults study. Int J Behav Nutr Phys Act. 2021 Sep 23;18(1):129. doi: 10.1186/s12966-021-01199-4. PMID 34556146
- [Result] McAvoy CR, Moore CC, Aguiar EJ, Ducharme SW, Schuna JM Jr, Barreira TV, Chase CJ, Gould ZR, Amalbert-Birriel MA, Chipkin SR, Staudenmayer J, Tudor-Locke C, Mora-Gonzalez J. Correction: Cadence (steps/min) and relative intensity in 21 to 60-year-olds: the CADENCE-adults study. Int J Behav Nutr Phys Act. 2022 Jun 2;19(1):62. doi: 10.1186/s12966-022-01295-z. No abstract available. PMID 35655283
- [Result] Mora-Gonzalez J, Gould ZR, Moore CC, Aguiar EJ, Ducharme SW, Schuna JM Jr, Barreira TV, Staudenmayer J, McAvoy CR, Boikova M, Miller TA, Tudor-Locke C. A catalog of validity indices for step counting wearable technologies during treadmill walking: the CADENCE-adults study. Int J Behav Nutr Phys Act. 2022 Sep 8;19(1):117. doi: 10.1186/s12966-022-01350-9. PMID 36076265
- [Result] Moore CC, Aguiar EJ, Ducharme SW, Tudor-Locke C. Development of a Cadence-based Metabolic Equation for Walking. Med Sci Sports Exerc. 2021 Jan;53(1):165-173. doi: 10.1249/MSS.0000000000002430. PMID 32555022
- [Result] Aguiar EJ, Gould ZR, Ducharme SW, Moore CC, McCullough AK, Tudor-Locke C. Cadence-based Classification of Minimally Moderate Intensity During Overground Walking in 21- to 40-Year-Old Adults. J Phys Act Health. 2019 Dec 1;16(12):1092-1097. doi: 10.1123/jpah.2019-0261. Epub 2019 Nov 6. PMID 31698337
- [Result] Ducharme SW, Lim J, Busa MA, Aguiar EJ, Moore CC, Schuna JM Jr, Barreira TV, Staudenmayer J, Chipkin SR, Tudor-Locke C. A Transparent Method for Step Detection using an Acceleration Threshold. J Meas Phys Behav. 2021 Dec;4(4):311-320. doi: 10.1123/jmpb.2021-0011. Epub 2021 Oct 25. PMID 36274923
- [Derived] McAvoy CR, Miller TA, Aguiar EJ, Ducharme SW, Moore CC, Schuna JM Jr, Barreira TV, Chase CJ, Gould ZR, Amalbert-Birriel MA, Chipkin SR, Staudenmayer J, Tudor-Locke C, Bucko A, Mora-Gonzalez J. Cadence (steps/min) and relative intensity in 61 to 85-year-olds: the CADENCE-Adults study. Int J Behav Nutr Phys Act. 2023 Nov 29;20(1):141. doi: 10.1186/s12966-023-01543-w. PMID 38031156
- [Derived] McAvoy CR, Moore CC, Aguiar EJ, Ducharme SW, Schuna JM Jr, Barreira TV, Chase CJ, Gould ZR, Amalbert-Birriel MA, Chipkin SR, Staudenmayer J, Tudor-Locke C, Mora-Gonzalez J. Cadence (steps/min) and relative intensity in 21 to 60-year-olds: the CADENCE-adults study. Int J Behav Nutr Phys Act. 2021 Feb 10;18(1):27. doi: 10.1186/s12966-021-01096-w. PMID 33568188